CLINICAL TRIAL: NCT00364832
Title: An Open-label, Multicenter, Randomized Study to Determine Dose Conversion Factors at Different Frequencies of Administration After Switching From Maintenance Treatment With Subcutaneous Epoetin Alfa or Beta to Maintenance Treatment With Subcutaneous RO0503821 in Dialysis Patients With Chronic Renal Anemia
Brief Title: A Study of Subcutaneous (sc) Mircera in Dialysis Patients With Chronic Renal Anemia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA16286
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Results first posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-10

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (9):
- Cohort A (0.4/150, 1x/ Week) (Experimental): Eligible participant will be administered RO0503821 (methoxy polyethylene glycol-epoetin beta [Mircera]) SC using a dose conversion factor of 0.4/150 microgram (mcg)/ kilogram (kg) of the previous weekly erythropoiesis stimulating agents (ESA) dose, (equal to 50% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants will be followed-up for two optional treatment extension periods (54 weeks each).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort B (0.4/150, 1x/ 3 Weeks) (Experimental): Eligible participant will be administered RO0503821 SC using a dose conversion factor of 0.4/150 mcg/kg of the previous weekly ESA dose, (equal to 50% assumed equi-effective dose) once every three weeks up to 19 weeks. After 19 weeks of core treatment period, participants will be followed-up for two optional treatment extension periods (54 weeks each).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort C (0.4/150, 1x/ 4 Weeks) (Experimental): Eligible participant will be administered RO0503821 SC using a dose conversion factor of 0.4/150 mcg/kg of the previous weekly ESA dose, (equal to 50% assumed equi-effective dose) once every four weeks up to 21 weeks. After 21 weeks of core treatment period, participants will be followed-up for two optional treatment extension periods (54 weeks each).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort D (0.8/150, 1x/ Week) (Experimental): Eligible participant will be administered RO0503821 SC using a dose conversion factor of 0.8/150 mcg/kg of the previous weekly ESA dose, (equal to 100% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants will be followed-up for two optional treatment extension periods (54 weeks each).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort E (0.8/150, 1x/ 3 Weeks) (Experimental): Eligible participant will be administered RO0503821 SC using a dose conversion factor of 0.8/150 mcg/kg of the previous weekly ESA dose, (equal to 100% assumed equi-effective dose) once every three weeks up to 19 weeks. After 19 weeks of core treatment period, participants will be followed-up for two optional treatment extension periods (54 weeks each).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort F (0.8/150, 1x/ 4 Weeks) (Experimental): Eligible participant will be administered RO0503821 SC using a dose conversion factor of 0.8/150 mcg/kg of the previous weekly ESA dose, (equal to 100% assumed equi-effective dose) once every four weeks up to 21 weeks. After 21 weeks of core treatment period, participants will be followed-up for two optional treatment extension periods (54 weeks each).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort G (1.2/150, 1x/ Week) (Experimental): Eligible participant will be administered RO0503821 SC using a dose conversion factor of 1.2/150 mcg/kg of the previous weekly ESA dose, (equal to 150% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants will be followed-up for two optional treatment extension periods (54 weeks each).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort H (1.2/150, 1x/ 3 Weeks) (Experimental): Eligible participant will be administered RO0503821 SC using a dose conversion factor of 1.2/150 mcg/kg of the previous weekly ESA dose, (equal to 150% assumed equi-effective dose) once every three weeks up to 19 weeks. After 19 weeks of core treatment period, participants will be followed-up for two optional treatment extension periods (54 weeks each).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort I (1.2/150, 1x/ 4 Weeks) (Experimental): Eligible participant will be administered RO0503821 SC using a dose conversion factor of 1.2/150 mcg/kg of the previous weekly ESA dose, (equal to 150% assumed equi-effective dose) once every four weeks up to 21 weeks. After 21 weeks of core treatment period, participants will be followed-up for two optional treatment extension periods (54 weeks each).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — Differing doses and frequencies of sc administration

SUMMARY:
This study will determine the appropriate dose and frequency of administration of sc Mircera maintenance therapy in dialysis patients with chronic renal anemia who were previously receiving sc epoetin alfa or beta. The anticipated time on study treatment is 3-12 months and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* chronic renal anemia;
* on dialysis (hemodialysis or peritoneal dialysis) therapy for at least 3 months;
* receiving sc epoetin alfa or beta for at least 3 months prior to the run-in period.

Exclusion Criteria:

* women who are pregnant, breastfeeding or using unreliable birth control methods;
* use of any investigational drug within 30 days preceding the run-in phase, or during the run-in or study treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2001-10; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- United States (6):
  - Los Angeles, California
  - San Jose, California
  - Boston, Massachusetts
  - Cleveland, Ohio
  - Houston, Texas
  - Morgantown, West Virginia
- Germany (4):
  - Berlin
  - Mannheim
  - Villingen-Schwenningen
  - Wiesloch
- Italy (8):
  - Bari
  - Bergamo
  - Lecco
  - Lodi
  - Milan
  - Modena
  - Pavia
  - Vicenza
- Spain (4):
  - Barcelona
  - Madrid
  - Málaga
  - Santander

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Locatelli F, Villa G, de Francisco AL, Albertazzi A, Adrogue HJ, Dougherty FC, Beyer U; BA16286 Study Investigators. Effect of a continuous erythropoietin receptor activator (C.E.R.A.) on stable haemoglobin in patients with CKD on dialysis: once monthly administration. Curr Med Res Opin. 2007 May;23(5):969-79. doi: 10.1185/030079907x182103. PMID 17519064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 137 participants were enrolled in this study conducted from 15 October 2001 to 7 July 2003 (core study period) and 19 September 2002 to 7 July 2005 (extension study period) at 22 centers (8 in Italy, 6 in the US, 4 in Germany, and 4 in Spain).
Groups:
- Cohort A (0.4/150, 1x/ Week): Eligible participants were administered RO0503821 (methoxy polyethylene glycol-epoetin beta [Mircera]) subcutaneous (SC) using a dose conversion factor of 0.4/150 microgram (mcg)/ kilogram (kg) of the previous weekly erythropoiesis stimulating agents (ESA) dose, (equal to 50% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort B (0.4/150, 1x/ 3 Weeks): Eligible participants were administered RO0503821 SC using a dose conversion factor of 0.4/150 mcg/kg of the previous weekly ESA dose, (equal to 50% assumed equi-effective dose) once every three weeks up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort C (0.4/150, 1x/ 4 Weeks): Eligible participants were administered RO0503821 SC using a dose conversion factor of 0.4/150 mcg/kg of the previous weekly ESA dose, (equal to 50% assumed equi-effective dose) once every four weeks up to 21 weeks. After 21 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort D (0.8/150, 1x/ Week): Eligible participants were administered RO0503821 SC using a dose conversion factor of 0.8/150 mcg/kg of the previous weekly ESA dose, (equal to 100% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort E (0.8/150, 1x/ 3 Weeks): Eligible participants were administered RO0503821 SC using a dose conversion factor of 0.8/150 mcg/kg of the previous weekly ESA dose, (equal to 100% assumed equi-effective dose) once every three weeks up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort F (0.8/150, 1x/ 4 Weeks): Eligible participants were administered RO0503821 SC using a dose conversion factor of 0.8/150 mcg/kg of the previous weekly ESA dose, (equal to 100% assumed equi-effective dose) once every four weeks up to 21 weeks. After 21 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort G (1.2/150, 1x/ Week): Eligible participants were administered RO0503821 SC using a dose conversion factor of 1.2/150 mcg/kg of the previous weekly ESA dose, (equal to 150% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort H (1.2/150, 1x/ 3 Weeks): Eligible participants were administered RO0503821 SC using a dose conversion factor of 1.2/150 mcg/kg of the previous weekly ESA dose, (equal to 150% assumed equi-effective dose) once every three weeks up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Cohort I (1.2/150, 1x/ 4 Weeks): Eligible participants were administered RO0503821 SC using a dose conversion factor of 1.2/150 mcg/kg of the previous weekly ESA dose, (equal to 150% assumed equi-effective dose) once every four weeks up to 21 weeks. After 21 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- RO0503821 (1x/ Week): Eligible participants were administered SC RO0503821 once weekly (1x/ week) using a dose conversion factor of 0.4/150-, 0.8/150-, and 1.2/150 mcg/kilogram of the previous weekly ESA dose in Cohort A, Cohort D, and Cohort G, respectively for 19 weeks. The ESA dose 50%, 100%, and 150% assumed equi-effective dose for dose conversion factors 0.4/150, 0.8/150 and 1.2/150, respectively. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- RO0503821 (1x/ 3 Weeks): Eligible participants were administered SC RO0503821 once every three weeks (1x/ 3 weeks) using a dose conversion factor of 0.4/150-, 0.8/150-, and 1.2/150 mcg/kg of the previous weekly ESA dose in Cohort B, Cohort E, and Cohort H, respectively for 19 weeks. The ESA dose 50%, 100%, and 150% assumed equi-effective dose for dose conversion factors 0.4/150, 0.8/150 and 1.2/150, respectively. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- RO0503821 (1x/ 4 Weeks): Eligible participants were administered SC RO0503821 once every four weeks (1x/ 4 weeks) using a dose conversion factor of 0.4/150-, 0.8/150-, and 1.2/150 mcg/kg of the previous weekly ESA dose in Cohort C, Cohort F, and Cohort I, respectively for 21 weeks. The ESA dose 50%, 100%, and 150% assumed equi-effective dose for dose conversion factors 0.4/150, 0.8/150 and 1.2/150, respectively. After 21 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
Period: Core Period
Arm/Group | Cohort A (0.4/150, 1x/ Week) | Cohort B (0.4/150, 1x/ 3 Weeks) | Cohort C (0.4/150, 1x/ 4 Weeks) | Cohort D (0.8/150, 1x/ Week) | Cohort E (0.8/150, 1x/ 3 Weeks) | Cohort F (0.8/150, 1x/ 4 Weeks) | Cohort G (1.2/150, 1x/ Week) | Cohort H (1.2/150, 1x/ 3 Weeks) | Cohort I (1.2/150, 1x/ 4 Weeks) | RO0503821 (1x/ Week) | RO0503821 (1x/ 3 Weeks) | RO0503821 (1x/ 4 Weeks)
Started | 16 | 15 | 15 | 16 | 16 | 12 | 16 | 15 | 16 | 0 | 0 | 0
Completed | 14 | 13 | 14 | 15 | 16 | 12 | 12 | 14 | 16 | 0 | 0 | 0
Not Completed | 2 | 2 | 1 | 1 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0
Not completed — Early Withdrawals | 2 | 2 | 1 | 1 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0
Period: Extension Year 1
Arm/Group | Cohort A (0.4/150, 1x/ Week) | Cohort B (0.4/150, 1x/ 3 Weeks) | Cohort C (0.4/150, 1x/ 4 Weeks) | Cohort D (0.8/150, 1x/ Week) | Cohort E (0.8/150, 1x/ 3 Weeks) | Cohort F (0.8/150, 1x/ 4 Weeks) | Cohort G (1.2/150, 1x/ Week) | Cohort H (1.2/150, 1x/ 3 Weeks) | Cohort I (1.2/150, 1x/ 4 Weeks) | RO0503821 (1x/ Week) | RO0503821 (1x/ 3 Weeks) | RO0503821 (1x/ 4 Weeks)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 (Participants (Cohorts A, D, and G) who completed core, entered extension period (entry optional).) | 17 (Participants (Cohorts B, E, and H) who completed core, entered extension period (entry optional).) | 27 (Participants (Cohorts C, F, and I) who completed core, entered extension period (entry optional).)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15 | 17
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 10
Not completed — Early Withdrawals | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 10
Period: Extension Year 2
Arm/Group | Cohort A (0.4/150, 1x/ Week) | Cohort B (0.4/150, 1x/ 3 Weeks) | Cohort C (0.4/150, 1x/ 4 Weeks) | Cohort D (0.8/150, 1x/ Week) | Cohort E (0.8/150, 1x/ 3 Weeks) | Cohort F (0.8/150, 1x/ 4 Weeks) | Cohort G (1.2/150, 1x/ Week) | Cohort H (1.2/150, 1x/ 3 Weeks) | Cohort I (1.2/150, 1x/ 4 Weeks) | RO0503821 (1x/ Week) | RO0503821 (1x/ 3 Weeks) | RO0503821 (1x/ 4 Weeks)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 14 (A portion of participants who completed Extension Year 1, entered Extension Year 2 (entry optional).) | 14 (A portion of participants who completed Extension Year 1, entered Extension Year 2 (entry optional).)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 3
Not completed — Early Withdrawals | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 3

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population was considered for analysis which included all randomized participants.
Groups:
- Cohort A (0.4/150, 1x/ Week): Eligible participants were administered RO0503821 SC using a dose conversion factor of 0.4/150 mcg/kg of the previous weekly ESA dose, (equal to 50% assumed equi-effective dose) once weekly up to 19 weeks. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- Total: Total of all reporting groups
Arm/Group | Cohort A (0.4/150, 1x/ Week) | Cohort B (0.4/150, 1x/ 3 Weeks) | Cohort C (0.4/150, 1x/ 4 Weeks) | Cohort D (0.8/150, 1x/ Week) | Cohort E (0.8/150, 1x/ 3 Weeks) | Cohort F (0.8/150, 1x/ 4 Weeks) | Cohort G (1.2/150, 1x/ Week) | Cohort H (1.2/150, 1x/ 3 Weeks) | Cohort I (1.2/150, 1x/ 4 Weeks) | Total
Number analyzed (Participants) | 16 | 15 | 15 | 16 | 16 | 12 | 16 | 15 | 16 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (13.03) | 65.6 (11.29) | 64.8 (10.28) | 61.8 (13.51) | 64.1 (12.83) | 67.3 (13.30) | 62.7 (13.74) | 58.9 (13.12) | 64.1 (13.34) | 63.9 (12.63)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 8 | 5 | 6 | 5 | 7 | 4 | 5 | 7 | 52
  Male | 11 | 7 | 10 | 10 | 11 | 5 | 12 | 10 | 9 | 85

OUTCOME MEASURES:

1. Primary Outcome: Median Change From Baseline in Hemoglobin Levels to End of Initial Treatment Under Constant Dosing Regimen
Description: Median change from Baseline in hemoglobin (Hb) levels to end of initial treatment (EOIT) under constant dosing regimen was reported. For ease of interpretation, all individual slope values were multiplied by 42 to give an estimate of change in Hb values over six weeks. Baseline (Day -28 to Day 1) Hb values was calculated as the mean of the screening assessment (SA) and run-in period (Week -2 and -1). For all participants, an EOIT value was calculated as the last observed Hb value before a dose change or blood transfusion. For participants without any dose adjustments or blood transfusion, the EOIT value was identical to the Week 19 (or Week 21) value.
Time Frame: From Baseline (Day -28 to Day 1) to EOIT (Week 19 or Week 21)
Population: The ITT population was considered for analysis which included all randomized participants.
Measure: Median (Inter-Quartile Range); unit: gram per deciliter
Arm/Group | Cohort A (0.4/150, 1x/ Week) | Cohort B (0.4/150, 1x/ 3 Weeks) | Cohort C (0.4/150, 1x/ 4 Weeks) | Cohort D (0.8/150, 1x/ Week) | Cohort E (0.8/150, 1x/ 3 Weeks) | Cohort F (0.8/150, 1x/ 4 Weeks) | Cohort G (1.2/150, 1x/ Week) | Cohort H (1.2/150, 1x/ 3 Weeks) | Cohort I (1.2/150, 1x/ 4 Weeks)
Number analyzed (Participants) | 16 | 15 | 15 | 16 | 16 | 12 | 16 | 15 | 16
gram per deciliter | -0.80 [-1.60 to -0.36] | -0.60 [-1.01 to -0.16] | -0.29 [-0.91 to -0.23] | 0.02 [-0.40 to 0.52] | -0.14 [-0.60 to 0.27] | -0.28 [-0.77 to 0.11] | 0.65 [0.12 to 1.57] | 0.33 [-0.11 to 1.14] | 0.22 [-0.09 to 1.02]
Statistical Analysis 1: Comparison: Cohort A (0.4/150, 1x/ Week) vs Cohort D (0.8/150, 1x/ Week) vs Cohort G (1.2/150, 1x/ Week); All cohorts with dosing frequency 1x/ week (0.4, 0.8 and 1.2 dose group); Test type: Superiority or Other; Estimated Conversion Factor 90% CI = 0.81, 90% CI 2-sided [0.73 to 0.90] — To analyze dose conversion factors (CF), 2nd regression (R) analysis was performed on 3 different CF dose groups, using the R slope estimates of Hb change over 6 weeks. Equi-effective CF was interpolated using value that gives an Hb change of zero
Statistical Analysis 2: Comparison: Cohort B (0.4/150, 1x/ 3 Weeks) vs Cohort E (0.8/150, 1x/ 3 Weeks) vs Cohort H (1.2/150, 1x/ 3 Weeks); All cohorts with dosing frequency 1x/ 3 weeks (0.4, 0.8 and 1.2 dose group); Test type: Superiority or Other; Estimated Conversion Factor 90% CI = 0.72, 90% CI 2-sided [0.55 to 0.86] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort C (0.4/150, 1x/ 4 Weeks) vs Cohort F (0.8/150, 1x/ 4 Weeks) vs Cohort I (1.2/150, 1x/ 4 Weeks); All cohorts with dosing frequency 1x/ 4 weeks (0.4, 0.8 and 1.2 dose group); Test type: Superiority or Other; Estimated Conversion Factor 90% CI = 0.93, 90% CI 2-sided [0.81 to 1.09] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Median Change From Baseline in Hematocrit Levels to End of Initial Treatment Under Constant Dosing Regimen
Description: Median change from Baseline in hematocrit (Hct) levels to end of initial treatment under constant dosing regimen was reported. Baseline (Day -28 to Day 1) Hct values was calculated as the mean of the SA and run-in period (Weeks -2 and -1). For all participants, an EOIT value was calculated as the last observed Hct value before a dose change or blood transfusion. For participants without any dose adjustments or blood transfusion, the EOIT value was identical to the Week 19 (or Week 21) value.
Time Frame: From Baseline (Day -28 to Day 1) to EOIT (Week 19 or Week 21)
Population: The ITT population was considered for analysis which included all randomized participants.
Measure: Median (Inter-Quartile Range); unit: Percentage of Hct
Arm/Group | Cohort A (0.4/150, 1x/ Week) | Cohort B (0.4/150, 1x/ 3 Weeks) | Cohort C (0.4/150, 1x/ 4 Weeks) | Cohort D (0.8/150, 1x/ Week) | Cohort E (0.8/150, 1x/ 3 Weeks) | Cohort F (0.8/150, 1x/ 4 Weeks) | Cohort G (1.2/150, 1x/ Week) | Cohort H (1.2/150, 1x/ 3 Weeks) | Cohort I (1.2/150, 1x/ 4 Weeks)
Number analyzed (Participants) | 16 | 15 | 15 | 16 | 16 | 12 | 16 | 15 | 16
Percentage of Hct | -2.45 [-6.33 to -0.83] | -1.95 [-3.28 to -0.34] | -0.93 [-2.56 to -0.63] | 0.25 [-1.25 to 1.36] | -0.37 [-1.67 to 1.02] | -0.75 [-2.23 to 0.35] | 2.25 [0.72 to 4.08] | 1.22 [-0.18 to 3.09] | 0.73 [-0.34 to 2.86]

3. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure and Diastolic Blood Pressure Before and After Dialysis
Description: Mean Change from Baseline in systolic blood pressure (SBP) and diastolic blood pressure (DBP) is calculated as the end of treatment values minus the Baseline value. Baseline (Day -28 to Day 1) value is the measurements taken at screening assessment and run-in period (Weeks -2 and -1).
Time Frame: From Baseline (Day -28 to Day 1) to Week 126
Population: The safety population was considered for analysis which included all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury
Arm/Group | Cohort A (0.4/150, 1x/ Week) | Cohort B (0.4/150, 1x/ 3 Weeks) | Cohort C (0.4/150, 1x/ 4 Weeks) | Cohort D (0.8/150, 1x/ Week) | Cohort E (0.8/150, 1x/ 3 Weeks) | Cohort F (0.8/150, 1x/ 4 Weeks) | Cohort G (1.2/150, 1x/ Week) | Cohort H (1.2/150, 1x/ 3 Weeks) | Cohort I (1.2/150, 1x/ 4 Weeks)
Number analyzed (Participants) | 16 | 15 | 15 | 16 | 16 | 12 | 16 | 15 | 16
Millimeters of Mercury
  SBP before dialysis | -1 (25.5) | 7 (15.5) | 2 (30.4) | -8 (18.1) | -4 (10.8) | -6 (20.3) | -2 (21.4) | 1 (18.6) | -7 (20)
  SBP after dialysis | 0 (24.4) | 10 (34.3) | 1 (26.9) | -4 (25.2) | 7 (17.1) | -5 (27.6) | 0 (25) | -1 (27.1) | -7 (18.2)
  DBP before dialysis | -1 (14.2) | 1 (9) | 3 (12.5) | -3 (11.4) | -2 (9.4) | 2 (12.9) | -3 (11.9) | -0 (11.4) | 1 (8.6)
  DBP after dialysis | -3 (14.6) | 4 (10.4) | -1 (12.9) | -3 (15.8) | 0 (11.1) | 2 (13.4) | -3 (12.2) | 5 (10.2) | -5 (10.3)

4. Secondary Outcome: Mean Change in Pulse Rate
Description: Mean change in pulse rate was reported.
Time Frame: Up to Week 126
Population: The safety population was considered for analysis which included all participants who received at least one dose of study drug. Participants with available data at the time of evaluation were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Cohort A (0.4/150, 1x/ Week) | Cohort B (0.4/150, 1x/ 3 Weeks) | Cohort C (0.4/150, 1x/ 4 Weeks) | Cohort D (0.8/150, 1x/ Week) | Cohort E (0.8/150, 1x/ 3 Weeks) | Cohort F (0.8/150, 1x/ 4 Weeks) | Cohort G (1.2/150, 1x/ Week) | Cohort H (1.2/150, 1x/ 3 Weeks) | Cohort I (1.2/150, 1x/ 4 Weeks)
Number analyzed (Participants) | 16 | 15 | 15 | 16 | 16 | 12 | 15 | 15 | 16
Beats per minute | -6 (8.8) | -2 (9.1) | 7 (9.1) | -1 (13.7) | -1 (7.7) | 2 (8.1) | 2 (9.9) | 0 (6.3) | 1 (9.1)

5. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: Participants with marked laboratory abnormalities were reported. Marked abnormality criteria: Serum glutamic oxaloacetic transaminase (SGOT); high >25 units per litre (U/L), albumin (low < 31 grams per litre [g/L]), total protein (< 60 g/L), phosphate (high >1.45 millimoles per litre [mmol/L]); Low <0.84 mmol/L), potassium (high >5 mmol/L; Low <3.5 mmol/L), platelets (low:<150×10^9/L), White blood cells ([WBCs]); high: 10.8×10^9/L and Low:4.3×10^9/L), basophils (high:>0.15×10^9/L), eosinophils (high:>0.70×10^9/L), lymphocytes (low:<1.50×10^9/L), and neutrophils (low:<1.83×10^9/L).
Time Frame: Up to Week 126
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Cohort A (0.4/150, 1x/ Week) | Cohort B (0.4/150, 1x/ 3 Weeks) | Cohort C (0.4/150, 1x/ 4 Weeks) | Cohort D (0.8/150, 1x/ Week) | Cohort E (0.8/150, 1x/ 3 Weeks) | Cohort F (0.8/150, 1x/ 4 Weeks) | Cohort G (1.2/150, 1x/ Week) | Cohort H (1.2/150, 1x/ 3 Weeks) | Cohort I (1.2/150, 1x/ 4 Weeks)
Number analyzed (Participants) | 16 | 15 | 15 | 16 | 16 | 12 | 16 | 15 | 16
Participants
  SGOT, High | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin, Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Total protein, Low | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0

6. Secondary Outcome: Number of Participants With Any Adverse Events, Any Serious Adverse Events, And Deaths
Description: An Adverse Events (AEs) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Serious Adverse Events (SAEs) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is a significant medical event in the investigator's judgment or requires intervention to prevent one or other of these outcomes. The study design tested 3 different starting dose conversion factors at 3 different dosing schedules during the core study period. As study drug doses can be modified continually over time all results for the two long term safety periods were displayed by dose schedule group only.
Time Frame: Up to Week 126
Population: as for outcome 3
Measure: Number; unit: Participants
Groups:
- RO0503821 (1x/ Week): Eligible participants were administered subcutaneous (SC) RO0503821 once weekly (1x/ week) using a dose conversion factor of 0.4/150-, 0.8/150-, and 1.2/150 microgram (mcg)/kilogram (kg) of the previous weekly erythropoiesis stimulating agents (ESA) dose in Cohort A, Cohort D, and Cohort G, respectively for 19 weeks. The ESA dose 50%, 100%, and 150% assumed equi-effective dose for dose conversion factors 0.4/150, 0.8/150 and 1.2/150, respectively. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- RO0503821 (1x/ 3 Weeks): Eligible participants were administered subcutaneous (SC) RO0503821 once every three weeks (1x/ 3 weeks) using a dose conversion factor of 0.4/150-, 0.8/150-, and 1.2/150 mcg/kg of the previous weekly ESA dose in Cohort B, Cohort E, and Cohort H, respectively for 19 weeks. The ESA dose 50%, 100%, and 150% assumed equi-effective dose for dose conversion factors 0.4/150, 0.8/150 and 1.2/150, respectively. After 19 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
- RO0503821 (1x/ 4 Weeks): Eligible participants were administered subcutaneous (SC) RO0503821 once every four weeks (1x/ 4 weeks) using a dose conversion factor of 0.4/150-, 0.8/150-, and 1.2/150 mcg/kg of the previous weekly ESA dose in Cohort C, Cohort F, and Cohort I, respectively for 21 weeks. The ESA dose 50%, 100%, and 150% assumed equi-effective dose for dose conversion factors 0.4/150, 0.8/150 and 1.2/150, respectively. After 21 weeks of core treatment period, participants were followed-up for two optional treatment extension periods (54 weeks each).
Arm/Group | RO0503821 (1x/ Week) | RO0503821 (1x/ 3 Weeks) | RO0503821 (1x/ 4 Weeks)
Number analyzed (Participants) | 48 | 46 | 43
Participants
  Any AEs | 44 | 33 | 40
  Any SAEs | 15 | 13 | 20
  Deaths | 7 | 4 | 10

ADVERSE EVENTS:
Time Frame: Up to Week 126
Description: SAEs and non-serious AEs are reported in safety analysis set, which consists of all participants who received at least one dose of study drug. The study design tested 3 different starting dose conversion factors at 3 different dosing schedules during the core study period. As study drug doses can be modified continually over time all results for the two long term safety periods were displayed by dose schedule group only.
Arm/Group | RO0503821 (1x/ Week) | RO0503821 (1x/ 3 Weeks) | RO0503821 (1x/ 4 Weeks)
Serious Adverse Events (participants affected / at risk) | 15/48 | 13/46 | 20/43
Other Adverse Events (participants affected / at risk) | 36/48 | 30/46 | 39/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (1x/ Week) (N=48) | RO0503821 (1x/ 3 Weeks) (N=46) | RO0503821 (1x/ 4 Weeks) (N=43)
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1 | 3
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 2 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 1
Central line infection (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Catheter sepsis (Infections and infestations) | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0
Peritoneal tuberculosis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 3 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 1
Catheter related complication (General disorders) | 0 | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 2
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 1
Arteriopathic disease (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Necrosis ischaemic (Vascular disorders) | 1 | 0 | 0
Peripheral occlusive disease (Vascular disorders) | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0
Vascular pseudoaneurysm (Vascular disorders) | 0 | 1 | 0
Venous stenosis (Vascular disorders) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Hyperparathyroidism Secondary (Endocrine disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cataract Operation (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (1x/ Week) (N=48) | RO0503821 (1x/ 3 Weeks) (N=46) | RO0503821 (1x/ 4 Weeks) (N=43)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 6 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 0 | 2
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Nasopharyngitis (Infections and infestations) | 8 | 4 | 8
Upper respiratory tract infection (Infections and infestations) | 2 | 5 | 3
Influenza (Infections and infestations) | 2 | 1 | 4
Bronchitis (Infections and infestations) | 1 | 3 | 1
Central line infection (Infections and infestations) | 3 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 3
Vomiting (Gastrointestinal disorders) | 5 | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 5
Nausea (Gastrointestinal disorders) | 4 | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 1
Hypotension (Vascular disorders) | 8 | 5 | 8
Hypertension (Vascular disorders) | 6 | 4 | 6
Procedural hypotension (Injury, poisoning and procedural complications) | 6 | 0 | 9
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3 | 3 | 4
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 3 | 1
Pyrexia (General disorders) | 3 | 3 | 5
Asthenia (General disorders) | 2 | 2 | 3
Oedema peripheral (General disorders) | 1 | 4 | 0
Influenza like illness (General disorders) | 1 | 0 | 3
Malaise (General disorders) | 3 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Headache (Nervous system disorders) | 4 | 6 | 4
Dizziness (Nervous system disorders) | 2 | 5 | 3
Carotid artery atheroma (Nervous system disorders) | 0 | 3 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 4 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 3
Atrial fibrillation (Cardiac disorders) | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.